CLINICAL TRIAL: NCT02891122
Title: The Influence of Duration of Fluid Abstinence on Hypotension During General Anaesthesia Induction for Traumatic Hip Surgery in the Elderly
Brief Title: Effect of the Duration of Preoperative Fasting on Hypotension Induced by General Anesthesia in the Elderly Person
Acronym: JEÛNE PREOP
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: JEÛNE PREOPERATOIRE
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Preoperative Fasting and Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to determine if prolonged fasting represents an independent risk factor for hypotension during induction of general anesthesia in the elderly.

DETAILED DESCRIPTION:
Preoperative fasting aims to reduce the risk of adverse events (eg, inhalation), but may be responsible for dehydration whose consequence is a major hypotension. This problem of hypotension is important because it (MAP <55 mmHg) is directly correlated to the occurrence of pejorative events on the cardiac and renal level and even more so that the duration of the hypotension is long.

ELIGIBILITY:
Inclusion Criteria:

* Risk Score anesthetic ASA I-III
* Patients ≥ 70 years
* Suffering from a femoral neck fracture to be treated surgically:

  * either through prosthesis,
  * either by intramedullary nailing (gamma nail)

Exclusion Criteria:

* Risk Score anesthetic ASA IV
* Patient on Angiotensin Converting Enzyme (ACE) inhibitors or ARBs (ARA2) within 10 hours before surgery
* Obesity (BMI> 35) or weight <40kg
* Need to make a rapid sequence induction
* Inability to achieve the femoral block (standardization of induction) or patient refusal with respect to the technique.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients hospitalized for fracture of the proximal femur requiring surgical treatment
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Follow-up of the variation of the Mean arterial pressure | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Lafère, Doctor, Principal Investigator — CHRU de Brest
Locations (1):
- CHRU de Brest, Brest, France